CLINICAL TRIAL: NCT02083029
Title: Vagal Nerve Stimulation Assessed by the Diving Reflex: An Investigation Into Mechanisms of Asthma Death
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Prof A H Morice, Head Cardiorespiratory Studies Hull York Medical School University of Hull Castle Hill Hospital Cottingham, Hull University Teaching Hospitals NHS Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CTU070813
Record Dates: First submitted 2014-03-03; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Asthma; Syncope
Keywords: Asthma; Death; Mechanism; Syncope; Dive reflex
MeSH Terms: conditions — Asthma; Syncope; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Syncopal Asthmatic (Experimental): All subject undergo simulated dive reflex, with 30s facial immersion and continuous HR and BP monitoring with Nexfin over a period of 6 minutes.
  Interventions: Procedure: Simulated dive reflex
- Non Syncopal Asthmatic (Experimental): All subject undergo simulated dive reflex, with 30s facial immersion and continuous HR and BP monitoring with Nexfin over a period of 6 minutes.
  Interventions: Procedure: Simulated dive reflex
- Normal Volunteers (Experimental): All subject undergo simulated dive reflex, with 30s facial immersion and continuous HR and BP monitoring with Nexfin over a period of 6 minutes.
  Interventions: Procedure: Simulated dive reflex

INTERVENTIONS:
Procedure: Simulated dive reflex — All subjects undergo simulated dive reflex, with 30s facial immersion and continuous HR and BP monitoring with Nexfin over a period of 6 minutes.

SUMMARY:
The investigators' hypothesis is that dysregulation of autonomic function, as revealed during a simulated dive reflex, may result in an attenuation of the heart rate response to a greater degree in asthmatics who collapse during exacerbations of asthma than that seen in healthy individuals and in asthmatics without a history of syncope. The investigators will test this by assessing autonomic function through a dive reflex protocol.

DETAILED DESCRIPTION:
Tests of autonomic function are notoriously difficult to evaluate. Here the investigators required a well validated test of the dynamic cardiovascular response to an abrupt stimulus and considered the diving reflex the most reliable and practical. In man, the diving reflex acts as a vestigial reflex aimed at conserving oxygen storage during apnoeic facial immersion. Facial immersion activates a vagally-induced bradycardia and a sympathetically activated alpha-adrenergic peripheral vasoconstriction and hypertension. There are two triggers of the diving reflex, facial immersion in water and breath hold, both of which can impact on heart rate attenuation. Facial immersion can be further delineated into exposure to cold, wetness and pressure.

ELIGIBILITY:
Inclusion Criteria:

* Syncopal Asthmatics: Asthmatic patients with a history of syncope during asthma exacerbations
* Normal Asthmatics: Asthmatic patients on BTS Step 3 treatment (LABA/ICS) with no history of syncope during exacerbations
* Normal volunteers: no history of airways disease or syncope

Exclusion Criteria:

* • Subjects who are pregnant, or have pacemakers in situ are excluded from this study.

  * Subjects with significant cardiovascular disease are excluded from this study.
  * Those who are non-English speakers and special groups (i.e. mentally ill, children under 16 years of age, and those suffering from dementia) will be excluded.
  * No test will be performed on any subject during an acute worsening of asthma or upper airway infection. If the subject has had an upper airway infection in the last three weeks. Another appointment should be made unless the subject is unwilling to come back, in which case testing should continue. The number of days elapsed since the end of the airway infection should be recorded.
  * If the subject smokes: citric acid or capsaicin challenges must be performed at least one hour after the last cigarette has been smoked.
  * Subjects taking beta-blockers and calcium antagonists will be excluded from this study. No beta agonists should be taken within 6 hours of starting this study.
  * If the subject has taken any over the counter (OTC) cough mixture within the last twelve hours: If the subject is willing to come back another time for challenge testing, another appointment should be made. If the subject is unwilling to return another time, testing should proceed and the medication used recorded.
  * If the subject has had any food or drink products containing caffeine or menthol within the last hour. If the subject is unwilling to wait for 1 hour before starting the test, the subject should return another time. If the subject is unwilling to return another time, testing should proceed and the medication used recorded.
  * If the participant is currently involved in research, or within 3 months of participation in any type of research, they will be excluded from this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in heart rate from baseline | 2 minutes prior to facial immersion in water and in 10 second epochs continuously until 3 minutes after facial immersion
  Nexfin and ECG monitoring continuously measuring subject heart rate during dive protocol, over a period of 6 minutes. Beat to beat data is converted into mean HR per 10-second epoch and compared to a baseline value for each subject.

SECONDARY OUTCOMES:
Change in blood pressure from baseline | 2 minutes before facial immersion and continuously throughout dive protocol, over a period of 6 minutes
  Nexfin monitoring continuously measuring subject blood pressure (systolic, diastolic and mean arterial pressure) during dive protocol, over a period of 6 minutes. Beat to beat data is converted into mean blood pressure values per 10-second epoch and compared to a baseline value for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Alyn Morice, MD, Principal Investigator — Head Cardiorespiratory Studies Hull York Medical School University of Hull Castle Hill Hospital Cottingham
Locations (1):
- Hull Clinical Trials Unit, Respiratory academic department, Cottingham, Yorkshire, United Kingdom

REFERENCES:
- [Derived] Morjaria JB, Rowland T, Tailor P, Hyder S, Wright CE, Hart SP, Morice AH. Autonomic dysregulation: a mechanism of asthma death. Eur Respir J. 2014 Nov;44(5):1357-60. doi: 10.1183/09031936.00076414. Epub 2014 Aug 19. No abstract available. PMID 25142490